CLINICAL TRIAL: NCT03862820
Title: The Use of Dynamic Ultrasound for Prediction of Adhesions in Women Undergoing Repeated Cesarean Section, an Observational Prospective Study
Brief Title: Dynamic Ultrasound for Prediction of Adhesion Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Haroun YOSEF, Lecturer, Assiut University
Other Study IDs: 1984
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: dynamic ultrasound — move abdomen with ultrasound probe to predict intraabdominal adhesions

SUMMARY:
1. To validate the use of dynamic ultrasound for prediction of adhesions in women undergoing repeated cesarean section.
2. To detect the interobserver and intraobserver reliability of this method

DETAILED DESCRIPTION:
INTRODUCTION Cesarean section is life saving procedure that involve extraction of the baby from the abdomen of the mother for numerous fetal and maternal indications The rate of cesarean section has been rising dramatically in the last decade reaching up to 32 % of birth in USA in 2014 . The rate of cesarean section in Assiut university in Egypt reached about 38% in 2011.

Cesearen section is associated with many intraoperative and postoperative early and late complications. Early complications includes hemorrhage bladder and bowel injuries, sepsis and postoperative illeus . Remote complications include the occurrence of intraperitoneal adhesions.The incidence of adhesions varies according to many factors includes the number of previous cesarean section, type of suture material, hemostasis but usually incidence of adhesions after cesarean is between 12 and 75 % .

The presence of adhesions in repeated cesarean section increases the surgical difficulty and the incidence of bladder and bowel injuries . Multidisciplinary team should evaluate these patients before surgery. Few studies used ultrasound to evaluate the presence of adhesions before operation . However they either used transvaaginal ultrasound which may not be available or used a small sample size which does not reflect the value of this tool accurately. In our study we are trying to use transabdominal ultrasound on large sample size to evaluate the use of dynamic ultrasound perioperative in predicting adhesions.

AIM OF THE STUDY

1. To validate the use of dynamic ultrasound for prediction of adhesions in women undergoing repeated cesarean section.
2. To detect the interobserver and intraobserver reliability of this method. PATIENTS AND METHODS

   * Study setting and population From February 2019 to February 2020, all women undergoing repeated cesarean section in both Assiut university hospital and El Eman hospital will be candidates for this study.
   * Study design The study will be blinded prospective observational study where investigator will perform ultrasound to recruited women before their elective cesarean section then the obstetrician who is blinded to the ultrasound results will be asked to fill a form postoperative to report the presence site and extent of adhesions.
   * Eligible participants Inclusion criteria Pregnant women in third trimester planned to undergo elective cesarean section ,

Exclusion criteria Primary elective cesarean section.

* Interventions Pregnant women planned to do elective cesarean section will be examined by two examiners senior resident and the assistant lecturer on duty using Medison ultrasound 5 MHZ abdominal convex probe. The probe is placed on the site of previous cesarean incision then moved from above downward and from side to side and we ask the patient to breathe deeply then we record the movement of anterior uterine wall against anterior abdominal wall where positive sliding sign if the uterus move freely and negative sliding sign if there is limited mobility. Elective cesarean is done by the obstetrician on duty as scheduled who is blind to the ultrasound results and then we ask him to report if adhesions are absent or present and if present site and type of adhesions and the difficulty of cesarean in a subjective score from 0 to 10. Preoperative and postoperative hemoglobin level will be measured as an indirect indicator for the difficulty of cesarean section.
* Sample size We need some work.
* Statistical Analysis The data will be collected and entered on Microsoft access data base to be analyzed using the Statistical Package for Social Science (SPSS Inc., Chicago, version 16). Sensitivity, specificity, negative and positive predictive value for the sliding sign will be measured
* Ethical aspect The study protocol will be submitted to Assiut medical school ethical board for approval. All participants will sign a written consent in the study after reading the patient information sheet or having it read for them if they cannot read or write. Confidentially of patient data will be secured in all stage of the study. Women who refuse participation in the study will not be affected by any mean regarding the quality of care in our service.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women in third trimester planned to undergo elective cesarean section

Exclusion Criteria:

Primary elective cesarean section.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women planned for elective repeated section
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
presence of abdominal adhesion intra operative | 1 year
  mobile uterus against uterine wall

CONTACTS AND LOCATIONS:
Overall Officials: Ali Yosef, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No